CLINICAL TRIAL: NCT00261456
Title: The IMPACT Study - Identification of Men With a Genetic Predisposition to ProstAte Cancer: Targeted Screening in Men at Higher Genetic Risk and Controls
Brief Title: The IMPACT Study - Identification of Men With a Genetic Predisposition to ProstAte Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other); Royal Marsden NHS Foundation Trust (Other); Ronald and Rita McAulay Foundation (Unknown); BRCA Research and Cure Alliance (Unknown)
Responsible Party: Sponsor
Other Study IDs: 05/MRE07/25; CCR2598 (Other: CCR)
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; BRCA Mutation; Mismatch Repair Gene Mutation; Genetic Predisposition to Disease
Keywords: Prostate cancer; BRCA1; BRCA2; prostate screening; PSA; prostate biopsy; Lynch Syndrome; Mismatch Repair Genes; MLH1; MSH2; MSH6
MeSH Terms: conditions — Prostatic Neoplasms; Genetic Predisposition to Disease; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Serum, Plasma, Urine, Prostate tissue.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- BRCA1/2 carriers: Carriers of a BRCA1 or BRCA2 mutation.
  Interventions: Diagnostic Test: PSA test; Procedure: Prostate Biopsy
- BRCA1/2 non Carriers: Do not carry a mutation in either the BRCA1 or 2 genes that has been found in other members of the family.
  Interventions: Diagnostic Test: PSA test; Procedure: Prostate Biopsy
- Mismatch Repair gene mutation carriers: Carriers of a MSH2, MSH6 or MLH1 mutation.
  Interventions: Diagnostic Test: PSA test; Procedure: Prostate Biopsy
- Mismatch Repair gene mutation non-carriers: Do not carry a mutation in either the MLH1, MSH2 or MSH6 genes that has been found in other members of the family.
  Interventions: Diagnostic Test: PSA test; Procedure: Prostate Biopsy

INTERVENTIONS:
Diagnostic Test: PSA test — Patients tested for their level of Prostate Specific Antigen.
Procedure: Prostate Biopsy — A Prostate biopsy is given as an option to the patient if their PSA level is raised or at the end of 5 years screening.

SUMMARY:
The IMPACT study is an international targeted prostate screening study of men at increased prostate cancer risk due to the presence of known pathogenic mutations in BRCA1 and BRCA2 genes and Mis-Match Repair genes (MLH1, MSH6, MSH2).

There are only approximately 150 men with a known BRCA1 or BRCA2 mutation in the UK. Research has shown that these men are at an increased risk of developing prostate cancer but more information is needed about the pathogenesis of prostate cancer in this defined group and the role of screening in these men. The study will offer annual PSA screening to these men to determine the incidence of prostate cancer in this group. The study will also look at new markers of early prostate cancer in this cohort.

The power calculations for this study are 850 carriers and 850 controls (age-matched men without BRCA1/2. Mis match repair mutations). It is therefore essential to gain international collaboration to meet the target of recruiting 850 men with these known mutations and a control group of 850 men who have tested negative for a known familial mutation.

DETAILED DESCRIPTION:
Prostate cancer is a significant public health problem. In the EU approximately 200,000 men are diagnosed annually with prostate cancer. There are 24,000 cases per year in England and Wales and 10,000 deaths. The incidence is increasing, even when screen-detected cancers are considered, and within the next few years it will become the most common cancer in UK men.

that an alteration in the breast cancer predisposition genes BRCA1 and BRCA2, may predispose to prostate cancer (PC) and this study will increase this evidence-base. There is some evidence, at least in BRCA2 carriers, that the prostate cancer in these men may be more aggressive and so earlier detection could theoretically reduce mortality. It has been reported that unaffected individuals from families with multiple cases of PC show an increased percentage of raised PSA levels, but the use of PSA level and its predictive value in healthy males with BRCA1/2 mutations has not been studied. If PSA were to be used as a screening tool in BRCA1/2 mutation carriers, we would need to gain a better understanding of the pathogenesis of PC in these men and determine whether they have a different baseline PSA profile compared with controls.

The high prevalence of hormone-dependent/secreting tumours such as breast, ovary and prostate in BRCA1/2 carriers suggests an important role of hormones and their receptors in the development of cancer. Androgens and androgen receptors are considered crucial elements in PC pathogenesis. Therefore male sex hormones will be measured to determine the hormone profile in BRCA1/2 carriers compared with a control group. There is strong evidence that BRCA1/2 play an important role in DNA repair and cell cycling. Therefore, we will investigate abnormalities of the metabolic processes in individuals with a BRCA1/2 mutation where cell cycling may be abnormal. Analysis of proteins (proteomics) and metabolites (metabonomics) are powerful approaches to identifying proteins and metabolites involved in cancer formation. The analysis of the proteins and metabolites will enable us to investigate the effect of the presence of a BRCA1/2 mutation and aid in the identification of new biomarkers for prostate cancer.

The target population is a group of 850 males who carry a known pathogenic mutation in the BRCA1/2 genes (500 BRCA1 and 350 BRCA2). These men will be recruited through genetics clinics across the UK and the world. A control group of men who have tested negative for a known pathogenic mutation that is running in their family will also be recruited through the genetics clinics.

All participants will be invited to attend annually for 5 years for an appointment lasting approximately 30 minutes during which they will discuss the study in detail before giving their written consent agreeing to participate. They will have a 50ml blood sample taken and be asked to provide a urine sample every year. They will also be required to complete a short family and medical history questionnaire. These appointments will either take place at the centre they are registered at, at the Royal Marsden Hospital, or in their own home depending on the arrangements made with the collaborating consultant and patient preference.

The PSA level of all participants will be measured locally. If PSA is >3.0ng/ml, a ten core prostatic biopsy will be offered, carried out by a consultant urologist. Ten biopsies will be used for diagnostic purposes, with two extra biopsy samples taken for research analysis with the patients fully informed written consent prior to the procedure being carried out. If any of the ten cores identify the presence of prostate cancer, they will receive treatment for this as advised by their local centre. The PSA will be quality controlled by batch testing at a reference lab. If the value locally was <3.0ng/ml but is >3ng/ml in the reference lab it will be remeasured locally.

If high grade Prostatic Intraepithelial Neoplasia (PIN) is detected or if the sample is inconclusive then a sextant biopsy repeated after 6 weeks will be recommended, in accordance with the ERSPC protocol. If atypical acini are detected then immediate biopsy will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Male carriers of a known pathogenic BRCA1/2 or Mismatch Repair gene mutations (MSH2, MSH6, MLH1) or men testing negative for a known BRCA1/2/ Mismatch repair mutation (MSH2, MSH6, MLH1) in their family
* Aged between 40-69 years old
* WHO performance status 0-2
* No previous history of prostate cancer
* No previous prostate biopsy for raised PSA
* Absence of any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule
* Fully informed, written consent according to ICH/EU GCP and national/local regulations before subject registration.

Exclusion Criteria:

* Previous cancer with terminal prognosis of less than 5 years
* Previous prostate cancer

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Person must have a prostate.
Study Population: Any patient that meets the eligibility criteria and maybe attending a genetics clinic at a number of international centres that have gone through ethical approval.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2005-03; Primary Completion 2030-02-28 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint (BRCA) | Through study completion, a minimum of 10 years follow up in participants.
  To determine the yearly incidence of screen-detected prostate cancer in BRCA1 and BRCA2 mutation carriers compared with the control population (predictive test negative for a known familial BRCA1/2 gene mutation). "
Primary Endpoint (Mismatch Repair/Lynch Cohort) | Through study completion, a minimum of 10 years follow up in participants.
  To determine the yearly incidence of screen-detected prostate cancer in mismatch repair gene mutation carriers compared with the control population (predictive test negative for a known familial MMR gene mutation).

SECONDARY OUTCOMES:
PSA threshold for prostate cancer detection | Through study completion, a minimum of 10 years follow up in participants.
  To determine age-specific PSA levels (ug/L) for cancer detection in mutation carriers versus controls from:
  i) a group of men who are age matched (+/- 5 years) and who have a negative predictive genetic test ii) two population based screening studies
Positive Predictive value of PSA level for prostate cancer detection | Through study completion, a minimum of 10 years follow up in participants.
  To determine the positive predictive value of PSA using a threshold of 3.0ug/L for the development of prostate cancer in mutation carriers using 5 or more years' annual follow up compared with the control populations
Cancer Pathology (BRCA) | Through study completion, a minimum of 10 years follow up in participants.
  To determine the stage and pathology at cancer diagnosis of screen-detected prostate cancer in BRCA1 and BRCA2 mutation carriers compared with the control population (predictive test negative for a known familial BRCA1/2 gene mutation).
Cancer Pathology (Mismatch Repair/Lynch Cohort) | Through study completion, a minimum of 10 years follow up in participants.
  To determine the stage and pathology at cancer diagnosis of screen-detected prostate cancer in mismatch repair gene mutation carriers compared with the control population (predictive test negative for a known familial MMR gene mutation).

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind A Eeles, FRCP FRCR, Principal Investigator — Institute of Cancer Research and Royal Marsden Hospital
Locations (1):
- Cancer Genetics Unit, Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data can be applied for via the Data Access Committee

REFERENCES:
- [Background] Tischkowitz M, Eeles R; IMPACT study: Identification of Men with genetic predisposition to Prostate Cancer and its Clinical Treatment collaborators. Mutations in BRCA1 and BRCA2 and predisposition to prostate cancer. Lancet. 2003 Jul 5;362(9377):80; author reply 80. doi: 10.1016/S0140-6736(03)13823-8. No abstract available. PMID 12853213
- [Background] Cremers RG, Eeles RA, Bancroft EK, Ringelberg-Borsboom J, Vasen HF, Van Asperen CJ; IMPACT Steering Committee; Schalken JA, Verhaegh GW, Kiemeney LA. The role of the prostate cancer gene 3 urine test in addition to serum prostate-specific antigen level in prostate cancer screening among breast cancer, early-onset gene mutation carriers. Urol Oncol. 2015 May;33(5):202.e19-28. doi: 10.1016/j.urolonc.2015.01.018. Epub 2015 Mar 5. PMID 25746941
- [Background] Killick E, Morgan R, Launchbury F, Bancroft E, Page E, Castro E, Kote-Jarai Z, Aprikian A, Blanco I, Clowes V, Domchek S, Douglas F, Eccles D, Evans DG, Harris M, Kirk J, Lam J, Lindeman G, Mitchell G, Pachter N, Selkirk C, Tucker K, Zgajnar J, Eeles R, Pandha H. Role of Engrailed-2 (EN2) as a prostate cancer detection biomarker in genetically high risk men. Sci Rep. 2013;3:2059. doi: 10.1038/srep02059. PMID 23792811
- [Background] Whitaker HC, Kote-Jarai Z, Ross-Adams H, Warren AY, Burge J, George A, Bancroft E, Jhavar S, Leongamornlert D, Tymrakiewicz M, Saunders E, Page E, Mitra A, Mitchell G, Lindeman GJ, Evans DG, Blanco I, Mercer C, Rubinstein WS, Clowes V, Douglas F, Hodgson S, Walker L, Donaldson A, Izatt L, Dorkins H, Male A, Tucker K, Stapleton A, Lam J, Kirk J, Lilja H, Easton D; IMPACT Study Steering Committee; IMPACT Study Collaborators; UK GPCS Collaborators; Cooper C, Eeles R, Neal DE. The rs10993994 risk allele for prostate cancer results in clinically relevant changes in microseminoprotein-beta expression in tissue and urine. PLoS One. 2010 Oct 13;5(10):e13363. doi: 10.1371/journal.pone.0013363. PMID 20967219
- [Background] Mikropoulos C, Selkirk CGH, Saya S, Bancroft E, Vertosick E, Dadaev T, Brendler C, Page E, Dias A, Evans DG, Rothwell J, Maehle L, Axcrona K, Richardson K, Eccles D, Jensen T, Osther PJ, van Asperen CJ, Vasen H, Kiemeney LA, Ringelberg J, Cybulski C, Wokolorczyk D, Hart R, Glover W, Lam J, Taylor L, Salinas M, Feliubadalo L, Oldenburg R, Cremers R, Verhaegh G, van Zelst-Stams WA, Oosterwijk JC, Cook J, Rosario DJ, Buys SS, Conner T, Domchek S, Powers J, Ausems MG, Teixeira MR, Maia S, Izatt L, Schmutzler R, Rhiem K, Foulkes WD, Boshari T, Davidson R, Ruijs M, Helderman-van den Enden AT, Andrews L, Walker L, Snape K, Henderson A, Jobson I, Lindeman GJ, Liljegren A, Harris M, Adank MA, Kirk J, Taylor A, Susman R, Chen-Shtoyerman R, Pachter N, Spigelman A, Side L, Zgajnar J, Mora J, Brewer C, Gadea N, Brady AF, Gallagher D, van Os T, Donaldson A, Stefansdottir V, Barwell J, James PA, Murphy D, Friedman E, Nicolai N, Greenhalgh L, Obeid E, Murthy V, Copakova L, McGrath J, Teo SH, Strom S, Kast K, Leongamornlert DA, Chamberlain A, Pope J, Newlin AC, Aaronson N, Ardern-Jones A, Bangma C, Castro E, Dearnaley D, Eyfjord J, Falconer A, Foster CS, Gronberg H, Hamdy FC, Johannsson O, Khoo V, Lubinski J, Grindedal EM, McKinley J, Shackleton K, Mitra AV, Moynihan C, Rennert G, Suri M, Tricker K; IMPACT study collaborators; Moss S, Kote-Jarai Z, Vickers A, Lilja H, Helfand BT, Eeles RA. Prostate-specific antigen velocity in a prospective prostate cancer screening study of men with genetic predisposition. Br J Cancer. 2018 Jan;118(2):266-276. doi: 10.1038/bjc.2017.429. Epub 2018 Jan 4. PMID 29301143
- [Background] Moynihan C, Bancroft EK, Mitra A, Ardern-Jones A, Castro E, Page EC, Eeles RA. Ambiguity in a masculine world: Being a BRCA1/2 mutation carrier and a man with prostate cancer. Psychooncology. 2017 Nov;26(11):1987-1993. doi: 10.1002/pon.4530. Epub 2017 Sep 18. PMID 28812325
- [Result] Mitra AV, Bancroft EK, Barbachano Y, Page EC, Foster CS, Jameson C, Mitchell G, Lindeman GJ, Stapleton A, Suthers G, Evans DG, Cruger D, Blanco I, Mercer C, Kirk J, Maehle L, Hodgson S, Walker L, Izatt L, Douglas F, Tucker K, Dorkins H, Clowes V, Male A, Donaldson A, Brewer C, Doherty R, Bulman B, Osther PJ, Salinas M, Eccles D, Axcrona K, Jobson I, Newcombe B, Cybulski C, Rubinstein WS, Buys S, Townshend S, Friedman E, Domchek S, Ramon Y Cajal T, Spigelman A, Teo SH, Nicolai N, Aaronson N, Ardern-Jones A, Bangma C, Dearnaley D, Eyfjord J, Falconer A, Gronberg H, Hamdy F, Johannsson O, Khoo V, Kote-Jarai Z, Lilja H, Lubinski J, Melia J, Moynihan C, Peock S, Rennert G, Schroder F, Sibley P, Suri M, Wilson P, Bignon YJ, Strom S, Tischkowitz M, Liljegren A, Ilencikova D, Abele A, Kyriacou K, van Asperen C, Kiemeney L; IMPACT Study Collaborators; Easton DF, Eeles RA. Targeted prostate cancer screening in men with mutations in BRCA1 and BRCA2 detects aggressive prostate cancer: preliminary analysis of the results of the IMPACT study. BJU Int. 2011 Jan;107(1):28-39. doi: 10.1111/j.1464-410X.2010.09648.x. Epub 2010 Sep 14. PMID 20840664
- [Result] Bancroft EK, Page EC, Castro E, Lilja H, Vickers A, Sjoberg D, Assel M, Foster CS, Mitchell G, Drew K, Maehle L, Axcrona K, Evans DG, Bulman B, Eccles D, McBride D, van Asperen C, Vasen H, Kiemeney LA, Ringelberg J, Cybulski C, Wokolorczyk D, Selkirk C, Hulick PJ, Bojesen A, Skytte AB, Lam J, Taylor L, Oldenburg R, Cremers R, Verhaegh G, van Zelst-Stams WA, Oosterwijk JC, Blanco I, Salinas M, Cook J, Rosario DJ, Buys S, Conner T, Ausems MG, Ong KR, Hoffman J, Domchek S, Powers J, Teixeira MR, Maia S, Foulkes WD, Taherian N, Ruijs M, Helderman-van den Enden AT, Izatt L, Davidson R, Adank MA, Walker L, Schmutzler R, Tucker K, Kirk J, Hodgson S, Harris M, Douglas F, Lindeman GJ, Zgajnar J, Tischkowitz M, Clowes VE, Susman R, Ramon y Cajal T, Patcher N, Gadea N, Spigelman A, van Os T, Liljegren A, Side L, Brewer C, Brady AF, Donaldson A, Stefansdottir V, Friedman E, Chen-Shtoyerman R, Amor DJ, Copakova L, Barwell J, Giri VN, Murthy V, Nicolai N, Teo SH, Greenhalgh L, Strom S, Henderson A, McGrath J, Gallagher D, Aaronson N, Ardern-Jones A, Bangma C, Dearnaley D, Costello P, Eyfjord J, Rothwell J, Falconer A, Gronberg H, Hamdy FC, Johannsson O, Khoo V, Kote-Jarai Z, Lubinski J, Axcrona U, Melia J, McKinley J, Mitra AV, Moynihan C, Rennert G, Suri M, Wilson P, Killick E; IMPACT Collaborators; Moss S, Eeles RA. Targeted prostate cancer screening in BRCA1 and BRCA2 mutation carriers: results from the initial screening round of the IMPACT study. Eur Urol. 2014 Sep;66(3):489-99. doi: 10.1016/j.eururo.2014.01.003. Epub 2014 Jan 15. PMID 24484606
- [Result] Page EC, Bancroft EK, Brook MN, Assel M, Hassan Al Battat M, Thomas S, Taylor N, Chamberlain A, Pope J, Raghallaigh HN, Evans DG, Rothwell J, Maehle L, Grindedal EM, James P, Mascarenhas L, McKinley J, Side L, Thomas T, van Asperen C, Vasen H, Kiemeney LA, Ringelberg J, Jensen TD, Osther PJS, Helfand BT, Genova E, Oldenburg RA, Cybulski C, Wokolorczyk D, Ong KR, Huber C, Lam J, Taylor L, Salinas M, Feliubadalo L, Oosterwijk JC, van Zelst-Stams W, Cook J, Rosario DJ, Domchek S, Powers J, Buys S, O'Toole K, Ausems MGEM, Schmutzler RK, Rhiem K, Izatt L, Tripathi V, Teixeira MR, Cardoso M, Foulkes WD, Aprikian A, van Randeraad H, Davidson R, Longmuir M, Ruijs MWG, Helderman van den Enden ATJM, Adank M, Williams R, Andrews L, Murphy DG, Halliday D, Walker L, Liljegren A, Carlsson S, Azzabi A, Jobson I, Morton C, Shackleton K, Snape K, Hanson H, Harris M, Tischkowitz M, Taylor A, Kirk J, Susman R, Chen-Shtoyerman R, Spigelman A, Pachter N, Ahmed M, Ramon Y Cajal T, Zgajnar J, Brewer C, Gadea N, Brady AF, van Os T, Gallagher D, Johannsson O, Donaldson A, Barwell J, Nicolai N, Friedman E, Obeid E, Greenhalgh L, Murthy V, Copakova L, Saya S, McGrath J, Cooke P, Ronlund K, Richardson K, Henderson A, Teo SH, Arun B, Kast K, Dias A, Aaronson NK, Ardern-Jones A, Bangma CH, Castro E, Dearnaley D, Eccles DM, Tricker K, Eyfjord J, Falconer A, Foster C, Gronberg H, Hamdy FC, Stefansdottir V, Khoo V, Lindeman GJ, Lubinski J, Axcrona K, Mikropoulos C, Mitra A, Moynihan C, Rennert G, Suri M, Wilson P, Dudderidge T; IMPACT Study Collaborators; Offman J, Kote-Jarai Z, Vickers A, Lilja H, Eeles RA. Interim Results from the IMPACT Study: Evidence for Prostate-specific Antigen Screening in BRCA2 Mutation Carriers. Eur Urol. 2019 Dec;76(6):831-842. doi: 10.1016/j.eururo.2019.08.019. Epub 2019 Sep 16. PMID 31537406
- [Result] Dias A, Brook MN, Bancroft EK, Page EC, Chamberlain A, Saya S, Amin J, Mikropoulos C, Taylor N, Myhill K, Thomas S, Saunders E, Dadaev T, Leongamornlert D, Dyrso Jensen T, Evans DG, Cybulski C, Liljegren A, Teo SH, Side L; IMPACT study collaborators and Steering Committee; Kote-Jarai Z, Eeles RA. Serum testosterone and prostate cancer in men with germline BRCA1/2 pathogenic variants. BJUI Compass. 2023 Jan 9;4(3):361-373. doi: 10.1002/bco2.156. eCollection 2023 May. PMID 37025481
- [Result] Bancroft EK, Page EC, Brook MN, Thomas S, Taylor N, Pope J, McHugh J, Jones AB, Karlsson Q, Merson S, Ong KR, Hoffman J, Huber C, Maehle L, Grindedal EM, Stormorken A, Evans DG, Rothwell J, Lalloo F, Brady AF, Bartlett M, Snape K, Hanson H, James P, McKinley J, Mascarenhas L, Syngal S, Ukaegbu C, Side L, Thomas T, Barwell J, Teixeira MR, Izatt L, Suri M, Macrae FA, Poplawski N, Chen-Shtoyerman R, Ahmed M, Musgrave H, Nicolai N, Greenhalgh L, Brewer C, Pachter N, Spigelman AD, Azzabi A, Helfand BT, Halliday D, Buys S, Ramon Y Cajal T, Donaldson A, Cooney KA, Harris M, McGrath J, Davidson R, Taylor A, Cooke P, Myhill K, Hogben M, Aaronson NK, Ardern-Jones A, Bangma CH, Castro E, Dearnaley D, Dias A, Dudderidge T, Eccles DM, Green K, Eyfjord J, Falconer A, Foster CS, Gronberg H, Hamdy FC, Johannsson O, Khoo V, Lilja H, Lindeman GJ, Lubinski J, Axcrona K, Mikropoulos C, Mitra AV, Moynihan C, Ni Raghallaigh H, Rennert G, Collier R; IMPACT Study Collaborators; Offman J, Kote-Jarai Z, Eeles RA. A prospective prostate cancer screening programme for men with pathogenic variants in mismatch repair genes (IMPACT): initial results from an international prospective study. Lancet Oncol. 2021 Nov;22(11):1618-1631. doi: 10.1016/S1470-2045(21)00522-2. Epub 2021 Oct 19. PMID 34678156
- [Result] Bancroft EK, Saya S, Page EC, Myhill K, Thomas S, Pope J, Chamberlain A, Hart R, Glover W, Cook J, Rosario DJ, Helfand BT, Hutten Selkirk C, Davidson R, Longmuir M, Eccles DM, Gadea N, Brewer C, Barwell J, Salinas M, Greenhalgh L, Tischkowitz M, Henderson A, Evans DG, Buys SS; IMPACT Study Steering Committee; IMPACT Collaborators; Eeles RA, Aaronson NK. Psychosocial impact of undergoing prostate cancer screening for men with BRCA1 or BRCA2 mutations. BJU Int. 2019 Feb;123(2):284-292. doi: 10.1111/bju.14412. Epub 2018 Jun 22. PMID 29802810
- [Result] Bancroft EK, Page EC, Brook MN, Pope J, Thomas S, Myhill K, Helfand BT, Talaty P, Ong KR, Douglas E, Cook J, Rosario DJ, Salinas M, Buys SS, Anson J, Davidson R, Longmuir M, Side L, Eccles DM, Tischkowitz M, Taylor A, Cruellas M, Ballestero EP, Cleaver R, Varughese M, Barwell J, LeButt M, Greenhalgh L, Hart R, Azzabi A, Jobson I, Cogley L, Evans DG, Rothwell J, Taylor N, Hogben M, Saya S; IMPACT Study Steering Committee; IMPACT Collaborators; Eeles RA, Aaronson NK. The psychosocial impact of prostate cancer screening for BRCA1 and BRCA2 carriers. BJU Int. 2024 Sep;134(3):484-500. doi: 10.1111/bju.16432. Epub 2024 Jun 5. PMID 38839570
- [Derived] Das S, Salami SS, Spratt DE, Kaffenberger SD, Jacobs MF, Morgan TM. Bringing Prostate Cancer Germline Genetics into Clinical Practice. J Urol. 2019 Aug;202(2):223-230. doi: 10.1097/JU.0000000000000137. Epub 2019 Jul 8. PMID 30730411
- See also: The IMPACT study website — http://impact.icr.ac.uk/
- See also: UK information point for eligible men — http://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-study-looking-at-screening-for-men-who-are-at-an-increased-risk-of-developing-prostate-cancer